CLINICAL TRIAL: NCT05829382
Title: A Randomized, Double-blind, Placebo Controlled, Cross-over Clinical Trial of Acute Safety and Biological Effects of a Polyphenol Supplement
Brief Title: A Study of Biological Effects of a Polyphenol Supplement
Acronym: MIDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MIDI
Record Dates: First submitted 2023-02-24; First posted 2023-04-25 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Healthy Aging

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo controlled, cross-over clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A randomized, double-blind, placebo controlled, cross-over trial to investigate the effect of the Investigational Product (DailyColors™) on age-related pathways in adults. Participants will receive DailyColors™ or placebo for a week, then one week wash-out, and then placebo/Dailycolors™ for a week, in random order. In addition, participants will be asked for consent to be contacted for participation in an open-label extension study for 3 months at a later date.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DailyColors™ group (Active Comparator): Capsules of 150 mg of the DailyColors™ blend
  The investigational product is a capsule containing 150mg of the following phytonutritients:
  Item Name Percent of Formula Apple Extract 10.0% Pomegranate Extract 10.0% Tomato Powder 2.5% Beet - Spray Dried 2.5% Olive Extract 7.5% Rosemary Extract 7.5% Green Coffee Bean Extract (C.A) 7.5% Kale - Freeze Dried 2.5% Onion Extract 10.0% Ginger Extract 10.0% Grapefruit Extract 2.5% Carrot - Air Dried 2.5% Grape Skin Extract 17.5% Blueberry Extract 2.5% Currant - Freeze Dried 2.5% Elderberry - Freeze Dried 2.5%
  Interventions: Dietary Supplement: DailyColors™
- Placebo group (Placebo Comparator): Micro crystalline cellulose will be used as the placebo, which will be produced with similar appearance as the active compound visually and regarding smell and taste.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: DailyColors™ — Capsule containing active ingredient administred daily by the participant during the trial period
  Arms: DailyColors™ group
Dietary Supplement: Placebo — Capsule containing placebo administered daily by the participant during the trial period
  Arms: Placebo group

SUMMARY:
A randomized, double-blind, placebo controlled, cross-over trial to investigate the effect of the Investigational Product "DailyColors™" (DC) on age-related pathways in adults.

The aim of this study is to measure the effects of acute treatment with DC on key pathways relevant to healthy ageing using blood biomarkers.

Based on power calculations a sample size of 20, is sufficient to detect an effect size of 0.46 at a power > 90%. To account for dropout the investigators will include 26 subjects in total.

DETAILED DESCRIPTION:
Aims:

The aim of this study is to measure the effects of acute treatment with DC on key pathways relevant to healthy ageing using blood biomarkers.

Hypotheses:

There will be preliminary evidence that the IP has positive clinical effects on biologically relevant pathways related to healthy aging of brain and muscle including blood markers of inflammation, oxidative stress markers, and trophic factors.

Design:

A randomized, double-blind, placebo controlled, cross-over trial to investigate the effect of the Investigational Product (DailyColors™) on age-related pathways in adults. Participants will receive DailyColors™ or placebo for a week, then one week wash-out, and then placebo/Dailycolors™ for a week, in random order. In addition, participants will be invited to participate in an open-label extension study for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, (NB Equal number of male and female participants)
* Age between 55 and 80
* Body Mass Index (BMI) over 25 (since this group is expected to have a some degree of inflammation and other metabolic changes and more likely to respond to the supplement)
* Willingness to complete questionnaires, records and diaries associated with the study and to complete all clinic visits
* Provided voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

* Alcohol or drug abuse in past year
* Subject has a known allergy to the test material's active or inactive ingredients
* Subjects with unstable, life-threatening medical conditions
* Use of polyphenol or phytochemical supplements
* Use of dietary supplements last month, except from cod liver oil or other vitamin D supplements
* Vegetarians and Vegans
* Clinically significant abnormal laboratory results at screening
* Participation in a clinical research trial within 30 days prior to randomization
* Individuals with dementia and/or who are unable to give informed consent
* Individuals with unusual high intake of fruit, berries, vegetable and/ or coffee intake, > 5 portions of fruit, berries and/or vegetables per day or > 5 cups of coffee per day
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Blood levels of CD38 | 3 weeks
  Change from baseline in the blood levels of CD38 at 1hour, 2 hours, 24 hours and week 1 and week 3. Blood CD38 is measured using commercially available immunoassays.
Blood levels of NAD+ | 3 weeks
  Change from baseline in the blood levels of NAD+ at 1hour, 2 hours, 24 hours and week 1 and 3. Blood NAD+ is measured using commercially available assay kits.

SECONDARY OUTCOMES:
Blood levels of biomarkers for inflammation | 3 weeks
  Change from baseline in the blood levels of inflammatory biomarkers, such as IL-6, TNF-α and IL-10, and IL-8 at week 1 and 3. All blood biomarkers are measured using commercially available immunoassays. All biomarkers have the same unit of measure, namely pg/mL.
Blood-based measurement of total antioxidant capacity | 3 weeks
  Change from baseline in the blood-based total antioxidant capacity at week 1 and 3, which are measured using commercially available assays.
Blood levels of 4-HNE | 3 weeks
  Change from baseline in the blood levels of 4-HNE at week 1 and week 3, which are measured using commercially available assays.
Blood levels of protein carbonyl | 3 weeks
  Change from baseline in the blood levels of protein carbonyl at week 1 and week 3, which are measured using commercially available assays.

CONTACTS AND LOCATIONS:
Overall Officials: Dag Aarsland, PhD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger Universitetssjukehus, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No